CLINICAL TRIAL: NCT07214168
Title: Factors That Affect Differential Switching and Patterns of ENDS Use Among Younger and Older Smokers: A Mixed Methods Approach
Brief Title: Vape Use Among Younger & Older Smokers
Acronym: ENDS
Status: Recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: The Center for Coordination of Analytics, Science, Enhancement and Logistics (CASEL) (Unknown); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Angela Aherrera, DrPH, MPH, Professor, Abramson Cancer Center at Penn Medicine
Other Study IDs: UPCC 13025; Protocol # 858558 (Other: UPenn IRB)
Record Dates: First submitted 2025-09-18; First posted 2025-10-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Smoking Cigarette; Smoking Behaviors; Vaping; Vaping Behaviors
Keywords: Vaping; Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking; Smoking; Vaping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine samples will be collected to analyze nicotine metabolites in the body, such as cotinine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to recruit 100 current cigarette smokers (50 young adults ages 21-34; 50 older adults ages 35-65) who have tried vaping or are currently vaping (dual users). The study will examine the trajectories in tobacco use (cigarettes and/or ENDS), including the nuanced differences in ENDS use (i.e., detailed device characteristics, user preferences, patterns of use), according to smoker age group.

ELIGIBILITY:
Inclusion Criteria:

* Male and female cigarette smokers who are between 21 and 65 years of age.
* Self-report having vaped at least once in the last six months (i.e. tried vaping) or are currently vaping.
* Self-report smoking at least 5 filtered cigarettes per week for at least the last 12 months.
* Not currently undergoing smoking cessation treatment or planning to quit prior to enrollment in the study.
* Able to attend 3 in-person visits in the Philadelphia area.
* Willing to smoke a cigarette in a ventilated smoking laboratory at each in-person visit.
* Capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form.
* Able to communicate fluently in English (i.e., speaking, writing, and reading).

Exclusion Criteria:

Smoking Behavior

-Use of any nicotine containing products other than cigarettes or ENDS. Participants reporting isolated use of other nicotine containing products less than 5 times per month are eligible to participate.

Alcohol and Drug Use

* History of substance abuse (other than nicotine) in the past 12 months and/or currently receiving medical treatment for substance abuse. Attendance at alcoholics anonymous or narcotics anonymous meetings will not be considered medical treatment for the purposes of this protocol.
* Current alcohol consumption that exceeds 25 standard drinks/week.

Medical

* Women, including all individuals assigned as female at birth, who are pregnant, breast feeding, or planning a pregnancy over the duration of the study period.
* Any psychiatric disorder that (as determined by the Principal Investigator) would interfere with study participation
* Serious or unstable medical condition. Applicable conditions will be evaluated on a case-by-case basis by the Principal Investigator.

General Exclusion

* Past, current, anticipated, or pending enrollment in another research program over the study period that could potentially impact participant safety, study data, and/or the study design as determined by the Principal Investigator.
* Any circumstance, medical condition, illness, disorder, adverse event (AE), or medication that could compromise participant safety or significantly impact study performance as determined by the Principal Investigator. Participants may be withdrawn for any of the aforementioned reasons at any point throughout the study.
* Significant non-compliance with the protocol and/or study design as determined by the Principal Investigator. Participants may be withdrawn at any point throughout the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Male and female cigarette smokers who are between 21 and 65 years of age.
  * Self-report having vaped at least once in the last six months (i.e. tried vaping) or are currently vaping.
  * Self-report smoking at least 5 filtered cigarettes per week for at least the last 12 months.
  * Able to attend 3 in-person visits in Philadelphia, PA
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Digital Diary (Mobile App) | 1 time per week for 5 months (Between Sessions)
  Participants will be asked to create an account for a mobile application that will serve as a digital diary to track any potential changes in tobacco product use, specifically ENDS and cigarette use, frequency of use for both products, and reasons for this change. The mobile app will ask the participant on a weekly basis whether there was any change to smoking and vaping habits from the past week. Collection of weekly data will provide granularity and a better understanding of the nuanced differences in ENDS use according to age group over the course of the 12-month enrollment period.
ENDS Use (Open Ended Response) | 5-6 months (at three time points)
  To identify the factors that impact ENDS use, participants will be asked to provide personal reasons to start vaping or try new ENDS products, continue vaping, or quit vaping.
ENDS Risk Beliefs | 5-6 months (at three time points)
  Participants will be asked questions adapted to ENDS use about their product perceptions, including measures of risk beliefs.
ENDS Perceived Health Risks | baseline
  Participants will be asked questions adapted to ENDS use about their product perceptions, including measures of perceived health risks.
ENDS Attitudes & Intentions | 5-6 months (at three time points)
  Participants will be asked to report on attitudes and intentions towards using ENDS, and social norms (the number of friends/family who smoke and/or vape and what friends/family behaviors/beliefs are on products; what the participants' beliefs about others approval of products are).
ENDS Personal Experience | 5-6 months (at three time points)
  Participants will be asked about personal experiences with ENDS use (physical sensation, experienced effects, ability to satisfy cravings, product problems, convenience of use, cost, regulation).

SECONDARY OUTCOMES:
Subjective Cigarette Ratings | 5-6 months (at three time points)
  Participants will provide subjective ratings of all cigarettes smoked during laboratory sessions using a 14-item, 100 mm visual analog scale (VAS) of cigarette characteristics (e.g., taste) used by the tobacco industry and our laboratory. Anchors are item-specific (e.g., taste: 0 = "very bad," 100 = "very good"), with lower scores indicating less favorable ratings. Subjective cigarette ratings will be assessed after each cigarette smoked in the laboratory across all sessions. The participant will also complete a modified version of the same form at each session for ENDS use. Participant ENDS subjective ratings will be collected after each vaping period in the laboratory (if applicable).
Puff Duration (via smoking topography) | 5-6 months (at three time points)
  Both smoking and vaping (if applicable) behaviors will be assessed using video-scored measures of topography (i.e., puffing behavior), which includes the number of puffs taken, and total inter-puff interval. A digital timestamp feature in opensource video editing software will be used to estimate start and end times for individual puffs based on various physical cues (i.e., inhaling, glowing cigarette tips or ENDS device).
Nicotine Metabolites (Urine Sample) | 5-6 months (at three time points)
  Spot urine samples will be collected using acid washed collection cups. Urine will be used to measure metals, aldehyde metabolites, cotinine, creatinine. Biospecimens will be frozen at < -80°C in freezers operated under a strict quality control system. The time in which each participant last vaped and when the biospecimen samples were collected will be recorded.
Carbon Monoxide (CO) assessment | 5-6 months (at three time points)
  CO levels will be measured using a breath CO monitor to assess tobacco exposure.The CO monitor is a handheld device that uses a disposable mouthpiece, reports CO in parts per million (ppm), and takes about 3 minutes to administer. Participants will smoke a cigarette of choice in the laboratory, and CO measurements will be collected to assess the difference before and after the cigarette smoked, or CO boost, to measure smoke exposure from a single cigarette. Collection of these secondary measures will allow the team to evaluate differences in tobacco and nicotine exposure between age groups, which may be impacted by participants' cigarette and ENDS product of choice and the potentially differing patterns of use between products.
Craving | 5-6 months (at three time points)
  Participants will report cigarette craving and nicotine withdrawal symptoms at the onset of each visit. Craving will be assessed using a summary score and two factor subscales (i.e., desire to smoke and craving due to anticipation of negative affect relief) from the 32-item Questionnaire on Smoking Urges (QSU).
Withdrawal | 5-6 months (at three time points)
  Withdrawal will be assessed using a summary score from the 20-item (21 items at Session 1 [D0]) revised version of the Withdrawal Symptom Checklist (WSC-W [1-week frame of reference]).
Attitude & Intention to Use Product | 5-6 months (at three time points)
  Participants' attitudes and intentions toward their cigarette packs will be assessed, similar to the lab's previous work on cigarette smoking that applied the Reasoned Action Approach. Likert-type semantic differential scales will be used (likely to use/not use, enjoyable/non enjoyable, harmful/not harmful). Participants will complete the Attitudes and Intentions Questionnaire across all sessions after smoking each lab cigarette. The participant will also complete a modified version of the same form at each session for ENDS use. Participant ENDS Attitudes & Intentions will be collected after each vaping period in the laboratory (if applicable).

CONTACTS AND LOCATIONS:
Overall Officials: Angela Aherrera, DrPH, MPH, Principal Investigator — University of Pennsylvania; Andrew Strasser, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Interdisciplinary Research on Nicotine Addiction, Philadelphia, Pennsylvania, United States